CLINICAL TRIAL: NCT05681169
Title: Schoolbased HPV-counselling and -Vaccination, a User-centred Intervention Targeting Children and Parents With Ethnic Minority Background
Brief Title: Schoolbased HPV-counselling and -Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus Municipality, Denmark (Other); Neighbourhood mothers, Gellerup (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Schoolbased HPV-vaccination
Record Dates: First submitted 2022-12-19; First posted 2023-01-12 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-06

CONDITIONS: HPV; Complex Intervention
Keywords: HPV; Vaccination program; Complex intervention; School-based; Patient involvement
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: Non-randomized implementation study, ratio between intervention and control group will be 1:4.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School-based HPV-counselling and HPV-vaccination (Experimental): 640 pupils
  Interventions: Other: School-based HPV-counselling and HPV-vaccination.
- Control group (No Intervention): The control population will be approximately 2560 children comparable in age and regions in Denmark with similar high concentration of ethnic minority populations.

INTERVENTIONS:
Other: School-based HPV-counselling and HPV-vaccination. — 1. Scholl-based parental HPV-counselling
  2. Scholl-based pupil HPV-counselling
  3. Scholl-based HPVV
  Arms: School-based HPV-counselling and HPV-vaccination

SUMMARY:
This study is designed as a non-randomized implementation study consisting of a user-centered school-based HPV-counselling and HPV-vaccination (HPVV) program. The aim is to improve HPVV coverage among children with ethnic minority background with minimum 10%-point in the intervention group.

DETAILED DESCRIPTION:
Background:

Human Papillomavirus (HPV)-related cancers are considered the most preventive cancer form due to vaccination. HPVV in Denmark is a part of a national children vaccination programme. Despite free access to vaccination, children and adolescents with ethnic minority background attend substantially less to the vaccination programme than native Danes (79 vs 93%). Among some ethnic minority groups, the HPVV coverage is as low as 65%. Barriers among ethnic minorities towards vaccination for HPV are complex, thus insufficient understanding of HPV, emotional barriers to sexuality and cultural taboos are of significance. Schoolbased vaccination can improve HPVV uptake, and counselling supporting vaccination could be significant when targeting ethnic minority families.

Aim:

To test schoolbased HPV-counselling of parents and pupils together with schoolbased HPVV, in schools with more than 25% ethnic minority pupils, to improve HPVV coverage among children with ethnic minority background.

Hypotheses and aims:

Hypothesis 1: It is possible to improve participation in HPVV in Denmark when combining HPV-counselling with school-based vaccination compared to general practitioner-based vaccination.

- Aim 1: To improve HPVV coverage among pupils attending schools with high concentration of non-native pupils. The investigators anticipate improving HPVV among ethnic minority pupils with at least 10%-point, and among native Danish pupils with at least 5%-point.

Hypothesis 2: It is possible to improve participation in HPVV among siblings to enrolled pupils, solely by improving HPV knowledge and awareness among their parents.

- Aim 2: To improve HPVV coverage among siblings to enrolled pupils.

Hypothesis 3: A close cooperation with user-representatives will improve feasibility and implementation.

- Aim 3: To develop and evaluate targeted counselling material concerning HPV and HPVV for parents and children with various ethnical backgrounds, eligible for national implementation.

Materials and methods:

Theoretical framework; The intervention is developed according to Complex Interventions Framework.Complex interventions contain several interacting components, and the guideline deals with development, assessment of feasibility, implementation, and evaluation. To operationalize the elements of the intervention, the investigators have applied a Logic Model, a graphic tool that illustrates the relationship between activities and intended outcome. By this, the investigators have combined theoretical knowledge and components of the intervention to accommodate to possible challenges in implementation.

Research design, study and control population; The intervention is conducted as a non-randomized implementation study. The intervention will be implemented schoolyear 2022/23. The intervention group consist of 640 children (11-13 years old) at 5 schools with > 25% ethnic minority pupils, located in Aarhus, Denmark. The control population will be approximately 2560 children comparable in age and regions with similar high concentration of ethnic minority populations.

Developed intervention;

The intervention consists of following core elements:

1. Scholl-based parental HPV-counselling
2. Scholl-based pupil HPV-counselling
3. Scholl-based HPVV

Counselling-material have been developed according to existing knowledge of communication to ethnic minority parents regarding health issues. The investigators have developed mainly video and animation, which also helps to ensure methodological rigor. All developed material has been validated and adapted in cooperation with users-representatives. To support implementation, the counselling process is designed to demand only few school-professional resources.

Parental counselling; A. Oral presentation (10 min) explaining HPV and HPVV. It will be given by a health professional (Medical doctor, Phd-student) at first school-parent meeting, with ethnic minority ambassadors present.

B. A simple printed presentation will be available in text and pictures (in Arabic, Turkish, Somali, English and Danish).

C. The oral presentation will be available as a video texted in Arabic, Turkish, Somali, English and Danish. It will be accessible in a Facebook-group, solely for parents included in the intervention.

To all parents not attending the school-parent meeting, the investigators will send all written material and opportunity to submit for participation to both an online personal mailbox and by letter with a stamped return-envelope.

Pupil counselling; A. In a school-nurse setting, it will consist of an animation (3 min), which illustrates facts about HPV and vaccination. The storytelling is a conversation between two kids, diverse in gender and ethnicity and contains subjects as nervousness.

B. The children will get a tote bag with a postcard, supporting the facts given in the animation and with an opportunity to submission by parents.

C. The school-nurse will facilitate a conversation about vaccination and nervousness, using 5 question-cards.

School-based HPVV; First vaccination (HPVV1) will be offered after element 1-2 have been completed; the second (HPVV2) will be offered minimum five months later. Both will be given at pre-defined dates during school hours by qualified doctors and nurses. Dates will be visible on posters at school and reminder will be send to parents via school communication platform and text messages if this is selected by parents when submitting their child for vaccination.

Evaluation plan:

Quantitative and qualitative outcome, see outcome section.

Power calculation; The investigators have enrolled 5 schools, corresponding to approximately 640 children. 2560 children will be allocated to the control group (1:4 ratio). In both groups, roughly half of these children will be native Danes and the other half will be ethnic minorities. Estimating that minority pupils have a HPVV coverage of 65%, the study will be able to detect a difference of approximately 10 percent points in vaccination coverage between intervention and control group in the stratified analyses with a risk of type 1 error of 5% and type 2 error of 10% (power 90%).

Data sources and statistical analysis; The intervention group has been identified by The Municipality of Aarhus and the control group will be identified in the Danish Civil Registration System, as will parents and siblings to both intervention and control groups. Information on children's' ethnicity, and demographic and socioeconomic status on parents will be obtained from Statistics Denmark. Data on HPVV 1 and 2 will be collected from The Danish National Health Service Register through the Danish Health Data Authority.

Demographic and socioeconomic characteristics will be presented as numbers and proportions and differences between intervention and control groups tested using Pearson's chi-squared test. Regression analyses will be used to estimate the relative risk of not being vaccinated between intervention and control group. If differences between intervention and control group are identified, both crude and adjusted estimates will be presented with 95% confidence intervals. All analyses will be performed using STATA V.17.

Ethical Considerations; The project will be conducted in accordance with the Good Clinical Practice Guidelines, and is reported to the Data Protection Agency in Central Denmark Region (ref.nr. 761330, 1-16-02-494-21) and Central Denmark Region's Committees on Biomedical Research (1-10-72-274-21). Parents must submit their child for vaccination via written informed consent. HPVV will be offered at pre-defined dates during school hours and provided by qualified medical professionals according to existing guidelines. Each HPVV will be registered in The National Danish Childhood Vaccination Register. All data will be handled according to the EU's General Data Protection Regulation and all sensitive information will be handled safely by using REDcap. The municipality of Aarhus will provide personal data on intervention group in order to perform the invention and data processing agreement about disclosure has been concluded. Interviews will be executed in accordance with the Helsinki Declaration's rules on voluntariness and anonymity.

Collaborators and user-representatives:

From the Municipality of Aarhus, Department of Children and Youth, we have a consultant dedicated to the project. The project has been approved by political and administrative leaders, and these are close collaborators. Two school-nurses are user-representatives. "Neighbourhood mothers" is a national volunteer organization of minority women trained in health, family and the Danish society. They constitute a large group of user-representatives. 10 mothers and children with various ethnic and social background are user-representatives, as well as 2 health professionals with cultural insight. The non-governmental organization "Sex og Samfund" [sex and society] has contributed with consultation regarding counselling material.

Perspectives:

The perspectives of initiating school-based HPVV, is to create equal opportunities for participation in primary prevention from HPV-related cancer for all children living in Denmark. Results from this study may be used in future preventive interventions, and material can be used in future school-based vaccination programs.

The investigators expect that the intervention will contribute to minimize misinformation and taboos related to HPVV among ethnic minority families, causing the intervention to indirectly benefit the HPVV attendance of the family's other children, and contribute to reduce inequality in Danish health care.

This project is the first step in a larger project with an overall aim to improve HPV-related cervical cancer prevention among minority groups in Denmark, which takes place in a cross regional collaboration between Aarhus University Hospital, Odense University Hospital and Randers Regional Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Pupils in 4th, 5th and 6th grade at 5 schools with > 25% ethnic minority pupils, located in Aarhus, Denmark.
* Age 9 - 15
* For vaccination there will be mandatory parental consent

Exclusion Criteria:

* Pupils from other schools or grades.
* Exclusion criteria from vaccination will be medical history of severe anaphylactic reaction
* Exclusion criteria from vaccination will be already initiated vaccination at general practitioner.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 640 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
HPV-vaccination coverage in intervention group | 1 year
  HPV coverage between intervention and control group as a total and stratified by ethnicity

SECONDARY OUTCOMES:
Estimated effect of HPV-counselling | 1 year
  HPVV coverage for siblings of included pupils compared to an age- and area matched control group.

OTHER OUTCOMES:
Qualitative perception of intervention | three months
  Parents' and school professionals' perceptions of the intervention will be qualitatively evaluated by focus-group interviews. The participants will be strategically selected among attending and non- attending, and represent various schools, cultural and socio-economic conditions. The interviews will be framed by a semi-structured interview guide, and data will be analysed and validated consecutively with Malterud's text analytical method

CONTACTS AND LOCATIONS:
Overall Officials: Lene K Seibæk, Prof, Study Chair — University of Aarhus
Locations (1):
- Anne Katrine Leonhard, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All of the results and experiences from the study are planned to be shared:
  * PhD-thesis with other researchers
  * Abstracts, posters and oral presentation at relevant conferences (EUROgin and IPVC (International Papillomavirus Conference) are planned)
  * Press and social media in Denmark
  * Oral presentations to organisations, the municipality of Aarhus and Neighbourhood Mothers.
  * Oral presentations to intervention interests, such as school nurses, teachers and school leaders.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available from spring 2023 to summer 2025.

REFERENCES:
- [Derived] Leonhard AK, Badre-Esfahani SK, Larsen MB, Petersen LK, Seibaek L. "Two shots for life. HPV-vaccination at your school". Co-creation of a complex intervention to reduce ethnic inequity in childhood HPV-vaccination in Denmark. PLoS One. 2025 Aug 20;20(8):e0323870. doi: 10.1371/journal.pone.0323870. eCollection 2025. PMID 40833975

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT05681169/Prot_SAP_000.pdf